CLINICAL TRIAL: NCT04195477
Title: Improving Health in Low Income Communities: Virtual Delivery of a Diabetes Prevention Program Facilitated With Community Care Coordination
Brief Title: vDPP Facilitated With Community Care Coordination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2000026747; U48DP006380-01-01 (Other: Centers for Disease Control and Prevention); U48DP006380-01 (NIH)
Record Dates: First submitted 2019-12-09; First posted 2019-12-12 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Diabetes Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- vDPP Full Study (Experimental): Participants will take part in a 52 week study receiving the vDPP intervention.
  Interventions: Behavioral: vDPP

INTERVENTIONS:
Behavioral: vDPP — virtual Diabetes Prevention Program

SUMMARY:
The goal of the proposed Implementation Research project is to assess the feasibility of and pathways for implementation of a virtually-delivered DPP (v-DPP) supported by community-based care coordination facilitated by community health workers (CHWs) and hospital-based community nurses (HCNs). The goal of the intervention is to improve body weight, blood pressure, diet quality, and physical activity levels among low-income individuals at risk for type 2 diabetes.

DETAILED DESCRIPTION:
Specific aims and hypotheses:

1. Conduct formative research with community partners (via focus groups and interviews with key stakeholders and a small pilot) to assess community, systemic, technology, and structural level barriers to implementation of a virtually-delivered Diabetes Prevention Program.

   Hypothesis: These efforts will identify individual and community needs, barriers, and resources affecting the feasibility of v-DPP implementation. In addition, strategies for facilitating the delivery of the v-DPP to low-income communities will be developed.
2. In collaboration with community partners, utilize strategies identified in Aim A1 to maximize impact of the v-DDP in target communities, as evidenced by measures of reach, effectiveness, adoption, implementation, and maintenance (RE-AIM) and assess factors influencing RE-AIM outcomes (e.g. social determinants of health, demographic variables, self-efficacy).

   Hypothesis: The v-DPP facilitated by community-based care coordination will produce favorable RE-AIM outcomes. Factors influencing these outcomes will be explored as well.
3. Demonstrate improvements in body weight, blood pressure, diet quality, and physical activity in low-income individuals at risk for type 2 diabetes who participate in a v-DPP facilitated by community-based care coordination.

   Hypothesis: The v-DPP, facilitated by community-based care coordination provided by CHWs and HCNs, will improve body weight, blood pressure, diet quality, and physical activity levels in the study communities.
4. Collaborate with community partners to develop and implement a strategic approach to sustain the v-DPP facilitated by community-based care coordination in the study communities and translate it to other community settings.

Hypothesis: The implementation approach will be packaged, including strategies for implementation in different settings and related costs, providing a process for implementation in other low-income communities in our region and nationally.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 25 kg/m2, based on self-reported weight and height;
* Eligible for Medicaid, as determined by self-reported income, household size, and Connecticut state guidelines for Medicaid eligibility;
* At risk for prediabetes, as evidenced by a score of 5 points or higher on the CDC prediabetes risk screening test. [https://www.cdc.gov/prediabetes/takethetest/]
* Participants in New Haven must also be residents of an ECC community (Housing Authority).
* Participants in Derby and Ansonia must demonstrate proof of residency of either town (i.e., bill or other mail addressed to them).

Exclusion Criteria:

* Failure to meet inclusion criteria;
* Anticipated inability to complete study protocol for any reason;
* Self-reported current eating disorder;
* Inability to exercise;
* Non-English speaking;
* Pregnant or planned pregnancy in next 12 months;
* Self-reported diagnosis of type 1 or type 2 diabetes;
* Failure to pass vDPP provider's required qualification step assessing readiness to change, when available.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2020-10-07 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Change in BMI | 16 weeks and 12 months
  Body mass index (BMI) will be measured as a participant's weight in kilograms divided by his/her height in meters squared. Height will be collected by a RA/CHW/HCN using a stadiometer at baseline and at 4 weeks.

SECONDARY OUTCOMES:
Change in Waist Circumference | 16 weeks and 12 months
  Waist circumference in centimeters will be collected at baseline and at 4 weeks.
Change in Total Cholesterol | 16 weeks and 12 months
  Total cholesterol (Tchol) will be collected at baseline and at 4 weeks.
Change in Triglycerides | 16 weeks and 12 months
  Triglycerides (TG) will be collected at baseline and at 4 weeks.
Change in High-density Lipoprotein | 16 weeks and 12 months
  High-density lipoprotein (HDL) will be collected at baseline and at 4 weeks.
Change in Diet Quality | 16 weeks and 12 months
  Dietary quality will be assessed at baseline and 4 weeks for the study. Participants will complete a 24-hour dietary recall using a web-based Automated Self-Administered 24-Hour Recall (ASA24) (available from the National Cancer Institute at ttp://riskfactor.cancer.gov/tools/instruments/asa24/), which will guide them through the process of completing the recall. Diet quality based on the information provided will be assessed using the Healthy Eating Index 2010 (HEI-2010).
Change in Physical Activity | 16 weeks and 12 months
  Physical activity level (PA) will be assessed at baseline and 4 weeks for the study. The International Physical Activity Questionnaire (IPAQ). It is a comprehensive tool containing information on weekly household and yard-work activities, occupational activity, transport, leisure time physical activity, and sedentary behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Perez-Escamilla, PhD, Principal Investigator — Professor of Public Health, Director of the Office of Public Health Practice, and Director of the Global Health Concentration at the Yale School of Public Health
Locations (2):
- United States (2):
  - Griffin Hospital, Derby, Connecticut
  - Yale University, New Haven, Connecticut

IPD SHARING:
Plan to Share IPD: No